CLINICAL TRIAL: NCT03396705
Title: Understanding the Molecular Basis of Normal Liver Regeneration
Brief Title: Liver Regeneration
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-5311
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Liver Diseases; Liver Cancer
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Liver Biopsy — liver tissue will be collected via core biopsy during liver resection surgery and post-operatively by fine needle aspiration biosy

SUMMARY:
The liver is the only visceral organ with a tremendous capacity to regenerate. We don't yet understand how normal liver regeneration occurs (on a molecular level) or how to distinguish between normal and "abnormal"/neoplastic regeneration. This study will characterize the role of the different liver cell types in the regeneration process and will examine gene expression changes in the various liver cell types.

DETAILED DESCRIPTION:
New studies are demonstrating that rodent models of the liver and liver disease are inadequate. The human liver is quite different and needs to be studied directly. The cell expression of human liver cells during regeneration has many implications for treatment of patients with cirrhosis and cancer.

This study will characterize the role of the different liver cell types in the regeneration process and will examine gene expression changes in the various liver cell types. We hypothesize that there is significant crosstalk among hepatocytes, macrophages, and T-cell subsets in the human liver, stimulating the regenerative process.

Tissue will be obtained from serial biopsies of "healthy" liver that is regenerating in patients who undergo liver resection for metastatic colorectal cancer. All participants must first provide written informed consent and meet study eligibility criteria. The first tissue sample will be collected intraoperatively, then serial fine-needle aspiration biopsies (FNAB) will be performed approx. 1 week following surgery, and 1 month following surgery. Liver regeneration will also be assessed using routine imaging of the liver at approx. 3 months.

Retrospective (previously collected diagnostic or biobanked) tissue is also being included for study, given lower than anticipated enrollment.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to provide written informed consent
* No history of liver disease or dysfunction

Exclusion Criteria:

* Patients who receive chemotherapy within the 6 weeks prior to their hepatectomy and/or would be started on active chemotherapy within the first 4 weeks post-hepatectomy.
* Patients requiring long-term anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing partial hepatectomy for colorectal cancer metastases, and meeting the eligibility criteria will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Gene expression | week 1 post-resection
  gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Mamatha Bhat, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No